CLINICAL TRIAL: NCT02833389
Title: A Phase Ib, Blinded, Randomized, Multicenter, Multiple-Ascending-Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of UTTR1147A Administered by Subcutaneous Injection in Patients With Non-Healing Neuropathic Diabetic Foot Ulcers
Brief Title: The Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of UTTR1147A in Participants With Neuropathic Non-Healing Diabetic Foot Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GX29915; 2015-003283-36 (EudraCT Number)
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Neuropathic Diabetic Foot Ulcers

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Cohort A - UTTR1147A, 0.8-6.0 cm^2, No Infection - Dose 1 (Experimental): Participants with 0.8-6.0 centimeters square (cm^2) index ulcer area at screening and no infection in index ulcer will receive UTTR1147A SC at Dose Level 1 for 12 weeks (a total of 4 doses).
  Interventions: Drug: UTTR1147A
- Cohort B - UTTR1147A, 0.8-6.0 cm^2, No Infection - Dose 2 (Experimental): Participants with 0.8-6.0 cm^2 index ulcer area at screening and no infection in index ulcer will receive UTTR1147A SC at Dose Level 2 for 12 weeks (a total of 4 doses).
  Interventions: Drug: UTTR1147A
- Cohort C - UTTR1147A, 0.8-6.0 cm^2, Mild Infection - Dose 2 (Experimental): Participants with 0.8-6.0 cm^2 index ulcer area at screening and mild infection in index ulcer will receive UTTR1147A SC at Dose Level 2 for 12 weeks (a total of 4 doses).
  Interventions: Drug: UTTR1147A
- Cohort D - UTTR1147A, 1.5-6.0 cm^2, Mild Infection - Dose 2 (Experimental): Participants with 1.5-6.0 cm^2 index ulcer area at screening and mild infection in index ulcer will receive UTTR1147A SC at Dose Level 2 for 12 weeks (a total of 4 doses).
  Interventions: Drug: UTTR1147A
- Cohort E - UTTR1147A, 0.8-6.0 cm^2, No infection - Dose 3 (Experimental): Participants with 0.8-6.0 cm^2 index ulcer area at screening and mild infection in index ulcer will receive UTTR1147A SC at Dose Level 3 for 12 weeks (a total of 4 doses).
  Interventions: Drug: UTTR1147A
- Placebo (Placebo Comparator): Participants will receive UTTR1147A matching placebo SC in each cohort for 12 weeks (a total of 4 doses).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — UTTR1147A matching placebo will be administered SC.
  Arms: Placebo
Drug: UTTR1147A — UTTR1147A will be administered SC.
  Other Names: RO7021610
  Arms: Cohort A - UTTR1147A, 0.8-6.0 cm^2, No Infection - Dose 1; Cohort B - UTTR1147A, 0.8-6.0 cm^2, No Infection - Dose 2; Cohort C - UTTR1147A, 0.8-6.0 cm^2, Mild Infection - Dose 2; Cohort D - UTTR1147A, 1.5-6.0 cm^2, Mild Infection - Dose 2; Cohort E - UTTR1147A, 0.8-6.0 cm^2, No infection - Dose 3

SUMMARY:
This trial will evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of repeat dosing of UTTR1147A in participants with neuropathic diabetic foot ulcers that do not respond adequately to standard wound care. Participants across multiple sites will be assigned to one of five cohorts (Cohort A, B, C, D, and E) based on the eligibility criteria and randomized to receive subcutaneous (SC) injections of either UTTR1147A or placebo over 12 weeks in addition to standard wound care.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Type 1 or Type 2 diabetes and confirmed peripheral neuropathy
* Have adequate circulation to the foot
* Have an ulcer area at screening up to 6 cm^2
* Up to date on all age-appropriate cancer screenings per local standards

Exclusion Criteria:

* Have current evidence of osteomyelitis, cellulitis, or evidence of systemic infection
* Have gangrene present on any part of the affected foot
* Known peripheral arterial disease requiring revascularization
* Have a glycated hemoglobin A1C level of greater than (>) 15% assessed at screening
* Are receiving oral or parenteral corticosteroids, immunosuppressive, or cytotoxic agents
* Have active malignancy or any history of a malignancy
* Use of oral antibiotics at the time of randomization for any reason in participants to be enrolled in Cohorts A, B, E, and any additional uninfected patient cohorts

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-11-14 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events | Baseline up to Day 141

SECONDARY OUTCOMES:
Percent Change from Baseline in Index Ulcer Surface Area at Weeks 6 and 12 | Baseline, Weeks 6 and 12
Percentage of Participants with Anti-Therapeutic (Anti-UTTR1147A) Antibodies | Day 1, 22, 64, 85, 99, early termination visit (up to Day 141)
Serum Concentration of UTTR1147A | Pre-dose (0 h) on Days 1, 22, 43, and 64, on Days 4, 8, 71, 85, and 99, early termination (up to Day 141)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (32):
- United States (10):
  - East Valley Foot and Ankle Specialists, Mesa, Arizona
  - Center for Clinical Research Inc.; i, San Francisco, California
  - Animas Foot and Ankle, Durango, Colorado
  - GF Professional Research Group Corporation, Miami Lakes, Florida
  - Podiatry 1st, Belleville, Illinois
  - Clinical Research Associates Of Central Pa , Llc, Altoona, Pennsylvania
  - Futuro Clinical Trials, McAllen, Texas
  - Endeavor Clinical Trials PA, San Antonio, Texas
  - 1Foot 2Foot Centre for Foot & Ankle Care PC, Suffolk, Virginia
  - Steven M. Waldman, SC, Wauwatosa, Wisconsin
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg
  - Bispebjerg Hospital, Copenhagen
  - Odense Universitetshospital; Endokrinologisk Afdeling, Odense
- Hungary (3):
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Semmelweis Egyetem, Budapest
  - Kenezy Korhaz Rendelointezet, Debrecen
- Italy (3):
  - Policlinico Universitario Campus Biomedico Di Roma; Farmacia, Rome, Lazio
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
- Spain (5):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Fundacion Hospital de Alcorcon, Alcorcón, Madrid
  - Hospital Universitario Cruces, Barakaldo, Vizcaya
  - Universidad Complutense de Madrid, Madrid
- United Kingdom (8):
  - Bradford Royal Infirmary, Bradford
  - Royal Derby Hospital; Medical School, Derby
  - Ipswich Hospital, Ipswich
  - St James University Hospital, Leeds
  - Kings College Hospital, London
  - University of East Anglia, Norfolk
  - Nottingham City Hospital, Nottingham
  - Northern General Hospital, Sheffield